CLINICAL TRIAL: NCT01726803
Title: Comparative Effectiveness of Management Strategies for Acute Low Back Pain
Brief Title: Comparative Effectiveness of Acute Low Back Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Julie Fritz, Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R18HS018672 (AHRQ)
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Primary Care; Physical Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Usual care arm will receive management as recommended by practice guidelines and directed by the primary care provider. The recommended stepped care approach is used with initial management of advice and education only and no referral to physical therapy during the initial 4 weeks.
  Interventions: Other: Usual Care
- Early Physical Therapy with Usual Care (Experimental): The Early Physical Therapy arm will receive the same advice and education intervention received by the usual care group and will be referred to receive 4 sessions of physical therapy during the first 4 weeks. The physical therapy protocol involves spinal manipulation and exercise.
  Interventions: Other: Early Physical Therapy with Usual Care; Other: Usual Care

INTERVENTIONS:
Other: Early Physical Therapy with Usual Care — The early physical therapy arm includes 4 total sessions. The first 2 sessions include use of thrust spinal manipulation with exercises for range of motion and strengthening of the spine. The final 2 sessions include the exercise component only.
  Arms: Early Physical Therapy with Usual Care
Other: Usual Care — The usual care intervention includes advice and education to remain active and provision of the Back Book highlighting these recommendations. Pharmaceuticals may be prescribed at the discretion of the primary care provider. Follow-up visits to primary care provided are recommended for all patients dissatisfied with their progress.

SUMMARY:
Current practice guidelines for patients with acute low back pain (LBP) recommend a stepped care approach with initial treatment of education and advice to remain active. Referral to physical therapy is considered only when patients fail to recover after a few weeks. Recent research has led to the identification a subgroup of patients likely to experience rapid, pronounced, and sustained decreases in disability and pain with a brief manipulation and exercise intervention, suggesting it may be more cost-effective to manage this sub-group with early referral to physical therapy instead of the usual care approach. The integration of this evidence into routine practice has not been evaluated. We will assess the outcomes of integrating this evidence into the management of patients with low back pain. The study is a randomized trial, comparing management with early manipulation with the current care process model. Patients fitting the inclusion criteria will be randomized into one of two groups. One group will be managed with the current care process model. The other group will be managed consistent with the decision rule recommending early referral for a brief manipulation and exercise intervention during the first 4 weeks. Patients will be followed over 1 year. Outcomes will include measures of disability, pain, satisfaction, and direct medical costs. The study will examine the costs and effectiveness of integrating the alternative care model into practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of pain and/or numbness between the 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the primary care provider, are originating from tissues of the lumbar region.
* Age 18 - 60 years
* Oswestry disability score > 20%
* Both of the following clinical decision rule criteria: a)Duration of current symptoms < 16 days; and b)Patient report of no symptoms (pain, numbness, etc.) distal to the knee in past 72 hours.

Exclusion Criteria:

* Prior surgery to the lumbosacral spine
* Any treatment for low back pain in past 6 months
* Current pregnancy
* Currently receiving treatment for LBP from another healthcare provider (e.g., chiropractic, massage therapy, injections, etc.)
* Presence of neurogenic LBP defined as the presence of either of the following:

  a) Positive ipsilateral or contralateral straight leg raise (reproduction of symptoms at <45 degrees); or b)Reflex, sensory, or strength deficits in a pattern consistent with lumbar nerve root compression
* Judgment of the primary care provider of "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, infection or systemic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PT, PhD, Principal Investigator — University of Utah and Intermountain Healthcare
Locations (2):
- United States (2):
  - Intermountain Health Care, Salt Lake City, Utah
  - The University of Utah Healthcare System, Salt Lake City, Utah

REFERENCES:
- [Derived] Sisco-Taylor BL, Magel JS, McFadden M, Greene T, Shen J, Fritz JM. Changes in Pain Catastrophizing and Fear-Avoidance Beliefs as Mediators of Early Physical Therapy on Disability and Pain in Acute Low-Back Pain: A Secondary Analysis of a Clinical Trial. Pain Med. 2022 May 30;23(6):1127-1137. doi: 10.1093/pm/pnab292. PMID 34613379
- [Derived] Magel J, Fritz JM, Greene T, Kjaer P, Marcus RL, Brennan GP. Outcomes of Patients With Acute Low Back Pain Stratified by the STarT Back Screening Tool: Secondary Analysis of a Randomized Trial. Phys Ther. 2017 Mar 1;97(3):330-337. doi: 10.2522/ptj.20160298. PMID 28204740
- [Derived] Fritz JM, Magel JS, McFadden M, Asche C, Thackeray A, Meier W, Brennan G. Early Physical Therapy vs Usual Care in Patients With Recent-Onset Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 13;314(14):1459-67. doi: 10.1001/jama.2015.11648. PMID 26461996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Early Physical Therapy With Usual Care
Started | 112 | 108
Completed | 105 | 107
Not Completed | 7 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Early Physical Therapy With Usual Care | Total
Number analyzed (Participants) | 112 | 108 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (10.2) | 38.3 (10.4) | 37.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 62 | 115
  Male | 59 | 46 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 99 | 103 | 202
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 2 | 3 | 5
  White | 90 | 89 | 179
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 112 | 108 | 220

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index
Description: 10-item Oswestry Disability Index assessing low back pain-related disability. Scores range from 0-100 with higher numbers indicating greater disability.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Usual Care: Usual care arm will receive management as recommended by practice guidelines and directed by the primary care provider. The recommended stepped care approach is used with initial management of advice and education only and no referral to physical therapy during the initial 4 weeks.
  Early Physical Therapy: The early physical therapy arm includes 4 total sessions. The first 2 sessions include use of thrust spinal manipulation with exercises for range of motion and strengthening of the spine. The final 2 sessions include the exercise component only.
  Usual Care: The usual care intervention includes advice and education to remain active and provision of the Back Book highlighting these recommendations. Pharmaceuticals may be prescribed at the discretion of the primary care provider. Follow-up visits to primary care provided are recommended for all patients dissatisfied with their progress.
- Early Physical Therapy: The Early Physical Therapy arm will receive the same advice and education intervention received by the usual care group and will be referred to receive 4 sessions of physical therapy during the first 4 weeks. The physical therapy protocol involves spinal manipulation and exercise.
  Usual Care: The usual care intervention includes advice and education to remain active and provision of the Back Book highlighting these recommendations. Pharmaceuticals may be prescribed at the discretion of the primary care provider. Follow-up visits to primary care provided are recommended for all patients dissatisfied with their progress.
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
units on a scale | 9.8 [7.9 to 11.7] | 6.6 [4.7 to 8.5]

2. Secondary Outcome: Numeric Pain Rating
Description: 0-10 numeric rating of low back pain intensity, score range from 0-10 with higher numbers indicating greater pain intensity.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
units on a scale | 1.8 [1.4 to 2.1] | 1.4 [1.1 to 1.7]

3. Secondary Outcome: EQ-5D
Description: European Quality of Life Measure, assesses general quality of life. Scores are expressed on a scale from 0 - 1.0 with higher scores representing greater quality of life.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
units on a scale | 0.88 [0.86 to 0.90] | 0.91 [0.88 to 0.93]

4. Secondary Outcome: Fear-Avoidance Beliefs Questionnaire (Work Subscale)
Description: Measures fear-avoidance beliefs related to work. Scores range from 0-42 with higher numbers representing greater levels of fear avoidance beliefs about work.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
units on a scale | 7.5 [6.2 to 8.8] | 5.2 [3.9 to 6.5]

5. Secondary Outcome: Patient Global Rating of Improvement (Percentage of Participants Reporting Successful Outcome)
Description: 15-point patient global rating scale. Patient is asked to rate current condition relative to condition at the beginning of treatment on a scale ranging from "A Very Great Deal Worse" to "A Very Great Deal Better". Higher numbers indicate greater self-rating. Those rating at least 12 are considered successful as a dichotomous outcome.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
percentage of participants | 49 | 64

6. Secondary Outcome: Health Care Utilization (MRI)
Description: Utilization of healthcare for low back pain (MRI utilization)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
participants | 3 | 4

7. Secondary Outcome: Pain Catastrophizing
Description: 13-item Pain Catastrophizing Scale assessing the extent of catastrophizing thinking is response to pain. Each item is scored 1-4 for a total score of 13-52. Higher numbers indicate greater levels of catastrophizing.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
units on a scale | 5.2 [4.0 to 6.4] | 3.0 [1.8 to 4.2]

8. Secondary Outcome: Lost Work Time
Description: Missed work due to LBP
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Usual Care | Early Physical Therapy
Number analyzed (Participants) | 112 | 108
participants | 46 | 40

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for physical therapy group after 4 weeks.
Arm/Group | Usual Care | Early Physical Therapy
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/108
Other Adverse Events (participants affected / at risk) | 0/112 | 13/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=112) | Early Physical Therapy (N=108)
side effects of physical therapy (Musculoskeletal and connective tissue disorders) | 0 | 13 — Patients reporting increased pain, spasm, stiffness, etc. following physical therapy treatment session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No